CLINICAL TRIAL: NCT05435807
Title: Investigation Of The Efficacy Of Therapeutic Neuroscience Education In Individuals With Fibromyalgia: A Randomized Controlled Trial
Brief Title: Therapeutic Neuroscience Education in Individuals With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Elif Gur Kabul, research assistant, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Neuroscience Education
Record Dates: First submitted 2022-06-18; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Clinical Pilates Exercises+TNE
  Interventions: Behavioral: Therapeutic Neuroscience Education
- control group (Experimental): Clinical Pilates Exercises
  Interventions: Behavioral: Therapeutic Neuroscience Education

INTERVENTIONS:
Behavioral: Therapeutic Neuroscience Education — Therapeutic Neuroscience Education (TNE) is an intervention used by physiotherapists, which can be defined as a cognitive behavioral therapy method. By helping patients better understand the biological process that underlies their painful condition, it aims to achieve therapeutic effects such as reducing pain and the fear associated with musculoskeletal injuries and increasing movement and functionality.

SUMMARY:
The aim of this study was to investigate the effects of Therapeutic Neuroscience Education (TNE) in individuals with Fibromyalgia (FM). The study included 25 females with FM, randomly separated into two groups as the intervention group (Clinical Pilates Exercises+TNE, n=11) and the control group (Clinical Pilates Exercises, n=14).

ELIGIBILITY:
Inclusion Criteria:

* age between 18-65 years,
* female gender,
* a VAS of at least 40mm to report the pain intensity of the last week,
* having been diagnosed with FM for at least 1 year to present a range of somatic and cognitive symptoms in addition to widespread pain,
* using a fixed dose of medication for at least the past 6 months (serotonin noradrenaline reuptake inhibitors [Ex, duloxetine, milnacipran]; alpha 2-delta receptor ligand [Ex, pregabalin]; gabapentinoids).

Exclusion Criteria:

* the presence of another disease which may affect the physical condition,
* cognitive impairment at a level preventing cooperation,
* being pregnant,
* inability to understand or speak Turkish,
* concurrent autoimmune or inflammatory disease,
* the presence of a central nervous system disease (eg multiple sclerosis, Parkinson's disease),
* serious psychiatric conditions (eg, psychotic disorders) that would prevent participation,
* participation in a rehabilitation program in the past year,
* have been exercising regularly for 6 months,
* not participating in at least 75% of treatments.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnare | 10 min
  Total score ranging from 0 to 100. Higher scores indicate worse functional status
Visual Analogue Scale | 5 min
  VAS is used to convert values that cannot be measured numerically, such as pain, into numerical values. Two end definitions of the parameter to be evaluated are written at the two ends of a 10 cm line and the patient is asked to mark this line indicating the appropriate level of their condition. In this study, 0='no pain' and 10='worst possible pain' were defined.
Widespread Pain Index | 10 min
  The WPI evaluates the patient's pain in the last week in terms of 19 regions and is scored between 0-19.
Symptom Severity Scale | 7 min
  The SSS is scored between 0-12.
Brief Pain Inventory | 7 min
  This is a short and easy-to-apply inventory that can be used to assess pain, which consists of the two sections of Pain Severity (4 items) and Pain Interference (7 items). The total score in both categories ranges from 0 to 10, with higher scores indicating more pain and more pain causes more disability.
Pain Catastrophizing Scale | 10 min
  The total score ranges from 0 to 52, with higher scores indicating a high level of catastrophizing.
Tampa Scale for Kinesiophobia | 10 min
  The total score ranges from 17 to 68, with a higher score indicating high kinesiophobia.

SECONDARY OUTCOMES:
Biopsychosocial Questionnaire | 10 min
  It includes 30 items that are answered using a 5-point Likert-type scale. Higher scores indicate a poor biopsychosocial status.
Dynamic Loewenstein Occupational Therapy Cognitive Assessment | 1 hour
  The DLOTCA battery has 28 subtests for 7 cognitive areas.Scoring consists of three components for each subtest:
  1. Before meditation score (5 points indicate the best performance).
  2. Mediation score (high score (4 or 5) indicates poor performance).
  3. After mediation score (5 points show the best performance).

CONTACTS AND LOCATIONS:
Overall Officials: Bilge Basakcı Calık, Prof., Principal Investigator — Pamukkale University; Ummuhan Bas ASLAN, Prof., Principal Investigator — Pamukkale University; Uğur Karasu, MD, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Merkezefendi, Turkey (Türkiye)